CLINICAL TRIAL: NCT03583398
Title: Health-related Quality of Life Following Transcatheter Aortic Valve Implantation Using Transaortic, Transfemoral Approaches and Surgical Aortic Valve Replacement - a Single-center Study
Brief Title: Health-related QoL Following TAVI TAo, TAVI TF and AVR
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Collaborators: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Principal Investigator, Aleksandra Stańska, MSc, Psychologist, Medical University of Gdansk
Other Study IDs: MUGdansk
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Quality of Life
Keywords: TAVI; quality of life; SAVR
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TAVI TAo
  Interventions: Procedure: transcatheter aortic valve implantation, surgical aortic valve replacement
- TAVI TF
  Interventions: Procedure: transcatheter aortic valve implantation, surgical aortic valve replacement
- AVR
  Interventions: Procedure: transcatheter aortic valve implantation, surgical aortic valve replacement

INTERVENTIONS:
Procedure: transcatheter aortic valve implantation, surgical aortic valve replacement — Transcatheter aortic valve implantation using transaortic and transfemoral access and surgical aortic valve replacement.

SUMMARY:
The aim of the study was to evaluate short- and long-term changes in QoL in patients undergoing TAVI and to assess differences in patient QoL when using the TAVI TAo approach compared with the transfemoral approach (TAVI TF) and surgical aortic valve replacement (SAVR).

ELIGIBILITY:
Inclusion Criteria:

* aortic valve stenosis

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elderly population with aortic valve stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life: EQ-5D-3L questionnaire | 1 month and 1 year follow-up
  EQ-5D-3L questionnaire

IPD SHARING:
Plan to Share IPD: No